CLINICAL TRIAL: NCT03263182
Title: Impact of the Safe Childbirth Checklist on Health Worker Childbirth Practices in Luapula Province of Zambia
Brief Title: Impact of the Safe Childbirth Checklist in Luapula Province of Zambia Province of Zambia
Status: Completed | Type: Observational
Sponsor: Clinton Health Access Initiative Inc. (Other)
Collaborators: Department for International Development, United Kingdom (Other Government); Ministry of Health, Zambia (Other Government)
Responsible Party: Sponsor
Other Study IDs: 3DE SCC
Record Dates: First submitted 2017-08-22; First posted 2017-08-28 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Maternal Death; Newborn Death
Keywords: childbirth; delivery
MeSH Terms: conditions — Maternal Death; Perinatal Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nchelenge Facilities: Purposively selected health facilities based on criteria including: high demand for services, perceived need for support for quality improvement, and presence of a SBA to mentor.
  Interventions: Behavioral: Introduction of the Safe Childbirth Checklist

INTERVENTIONS:
Behavioral: Introduction of the Safe Childbirth Checklist — 1. Adaptation of the SCC tool to Zambia: In order to produce a tool that is fully relevant to the Zambian context, a team of clinical experts from the MOH adapted the language of the SCC.
  2. Training of trainers on the SCC by international experts: Ariadne Labs has designed a training-of-trainers (TOT) for coach training to support quality improvement initiatives, including the implementation of the WHO SCC. Members of the district mentorship team for Nchelenge District will receive this type of TOT training.
  3. Following the TOT session, the district mentorship team will conduct facility-level training for health workers on using the SCC. Within target facilities, all public sector health workers will be invited to participate in the training.
  4. Mentorship and support to facility-level health workers on using the SCC: The district mentorship team will carry out coaching and support visits to health facilities following the initial SCC training.

SUMMARY:
This study would like to determine if the introduction of the Safe Childbirth Checklist and associated mentorship can improve the adherence of skilled birth attendants (SBAs) to the essential practices of childbirth delivery.

DETAILED DESCRIPTION:
This study will use a pre-post study design to measure health worker adherence to the essential practices for delivery care outlined in the Safe Childbirth Checklist (SCC). The intervention, including the introduction of the SCC and mentorship visits to support uptake, will be tested in four purposively selected health facilities in Nchelenge District, Luapula Province of Zambia. Since the essential delivery care practices outlined in the SCC are evidence-based practices broadly accepted to support positive clinical outcomes for mothers and infants, this evaluation will focus on adherence to the checklist rather than on patient outcomes. Data will be collected through observations of skilled birth attendants assisting with childbirth delivery before the start of the intervention and again at 3 months and 6 months post-intervention. A health worker questionnaire will be administered at the time that the SCC is introduced and six months later to gather their perspectives on incorporating the SCC into clinical practice in Zambia.

ELIGIBILITY:
Inclusion Criteria:

* For facility observations, all consecutive deliveries will be observed. If a pregnant woman or health worker declines to participate in the consent process, no observations will be recorded.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All births will be observed at any time of the day (with two data collectors taking 12-hour shifts). Observations will be conducted for a minimum of three days in all four facilities, or as long as required to observe at least 7 births. It may not be possible for the observer to observe every delivery process at all times, particularly if multiple observations are taking place at one time, so observations will relate to activities at four specific periods (pause points): on admission, when the mother starts pushing, through the delivery to one hour after delivery, and before discharge.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Change in the average proportion of observed, SCC tasks completed per birth from selected task list | Through study completion, an average of 6 months
  Numerator: Count of SCC tasks observed and completed for each delivery, according to the specifications for data collection outlined in the data collection procedures Denominator: Count of potential SCC items observed

SECONDARY OUTCOMES:
Characteristics of health workers participating in facility-level SCC training | Baseline
  Questionnaire to understand Health worker cadre and training
Feedback of health workers participating in facility-level SCC training | Baseline
  Proportion of health workers agreeing with statements on the clarity of the training and their confidence in using the SCC after the training
Feedback of health workers in participating facilities on SCC implementation | 6 months
  Questionnaire to understand Health worker cadre and training
Feedback of health workers in participating facilities on SCC implementation | 6 months
  Proportion of health workers agreeing with on ease of using the SCC and challenges faced in implementation

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Mudhune, Principal Investigator — Clinton Health Access Initiative, Nigeria; Francis Bwalya, Principal Investigator — Ministry of Health, Zambia
Locations (4):
- Zambia (4):
  - Kabuta Rural Health Centre, Nchelenge
  - Kambwali Rural Health Center, Nchelenge
  - Kashikishi Rural Health Centre, Nchelenge
  - St Paul's Mission Hospital, Nchelenge

IPD SHARING:
Plan to Share IPD: Undecided
This is yet to be finalized with the Ministry of Health, Zambia.

REFERENCES:
- [Background] Albolinoa S, Daglianaa G, et al. Safety and quality of maternal and neonatal pathway: A pilot study on the childbirth checklist in 9 Italian hospitals. Procedia Manufacturing. 2015; (3):242-249.
- [Background] Ariadne Labs. Implementing Checklists for Quality Improvement: The Namibian Experience using the WHO Safe Childbirth Checklist.
- [Background] Central Statistical Office (CSO), Ministry of Health (MOH), Tropical Diseases Research Centre (TDRC), University of Zambia, and Macro International Inc. (2014). Zambia Demographic and Health Survey 2014. Calverton, Maryland, USA: CSO and Macro International Inc.
- [Background] Davoodi R, Soltanifar A, et al. Efficacy of Evidence Based Care on Care Quality of Mother and Infant in 3 Teaching Hospitals: A Protocol. Patient Safety and Quality Improvement Journal. 2013 Dec 14; 2(2):97-100.
- [Background] Hayes RJ, Bennett S. Simple sample size calculation for cluster-randomized trials. Int J Epidemiol. 1999 Apr;28(2):319-26. doi: 10.1093/ije/28.2.319. PMID 10342698
- [Background] Haynes AB, Weiser TG, Berry WR, Lipsitz SR, Breizat AH, Dellinger EP, Herbosa T, Joseph S, Kibatala PL, Lapitan MC, Merry AF, Moorthy K, Reznick RK, Taylor B, Gawande AA; Safe Surgery Saves Lives Study Group. A surgical safety checklist to reduce morbidity and mortality in a global population. N Engl J Med. 2009 Jan 29;360(5):491-9. doi: 10.1056/NEJMsa0810119. Epub 2009 Jan 14. PMID 19144931
- [Background] Hirschhorn LR, Semrau K, Kodkany B, Churchill R, Kapoor A, Spector J, Ringer S, Firestone R, Kumar V, Gawande A. Learning before leaping: integration of an adaptive study design process prior to initiation of BetterBirth, a large-scale randomized controlled trial in Uttar Pradesh, India. Implement Sci. 2015 Aug 14;10:117. doi: 10.1186/s13012-015-0309-y. PMID 26271331
- [Background] Kumar S, Yadav V, Balasubramaniam S, Jain Y, Joshi CS, Saran K, Sood B. Effectiveness of the WHO SCC on improving adherence to essential practices during childbirth, in resource constrained settings. BMC Pregnancy Childbirth. 2016 Nov 8;16(1):345. doi: 10.1186/s12884-016-1139-x. PMID 27825321
- [Background] Kumari S, Panicker R, et al. Evaluation of the Safe Childbirth Checklist Program in Rajasthan, India: The How and What of the Evaluation Efforts. Journal of Public Health in Developing Countries. 2016 Aug 11;2(2);212-222.
- [Background] McCambridge J, Witton J, Elbourne DR. Systematic review of the Hawthorne effect: new concepts are needed to study research participation effects. J Clin Epidemiol. 2014 Mar;67(3):267-77. doi: 10.1016/j.jclinepi.2013.08.015. Epub 2013 Nov 22. PMID 24275499
- [Background] Moyer CA, Mustafa A. Drivers and deterrents of facility delivery in sub-Saharan Africa: a systematic review. Reprod Health. 2013 Aug 20;10:40. doi: 10.1186/1742-4755-10-40. PMID 23962135
- [Background] Ministry of Health [Zambia]. Health Sector Payroll Data. January 2014.
- [Background] Ministry of Health [Zambia]. Emergency Obstetric and Newborn Care (EmONC) Training Process Evaluation Report. February 2017.
- [Background] Ministry of Health [Zambia]. Zambia National Emergency Obstetric and Newborn Care (EmONC) Needs Assessment 2014-5. January 2017.
- [Background] Patabendige M, Senanayake H. Implementation of the WHO safe childbirth checklist program at a tertiary care setting in Sri Lanka: a developing country experience. BMC Pregnancy Childbirth. 2015 Feb 4;15:12. doi: 10.1186/s12884-015-0436-0. PMID 25648543
- [Background] Paxton A, Maine D, Freedman L, Fry D, Lobis S. The evidence for emergency obstetric care. Int J Gynaecol Obstet. 2005 Feb;88(2):181-93. doi: 10.1016/j.ijgo.2004.11.026. Epub 2005 Jan 8. PMID 15694106
- [Background] Spector JM, Agrawal P, Kodkany B, Lipsitz S, Lashoher A, Dziekan G, Bahl R, Merialdi M, Mathai M, Lemer C, Gawande A. Improving quality of care for maternal and newborn health: prospective pilot study of the WHO safe childbirth checklist program. PLoS One. 2012;7(5):e35151. doi: 10.1371/journal.pone.0035151. Epub 2012 May 16. PMID 22615733
- [Background] Spector JM, Lashoher A, Agrawal P, Lemer C, Dziekan G, Bahl R, Mathai M, Merialdi M, Berry W, Gawande AA. Designing the WHO Safe Childbirth Checklist program to improve quality of care at childbirth. Int J Gynaecol Obstet. 2013 Aug;122(2):164-8. doi: 10.1016/j.ijgo.2013.03.022. Epub 2013 Jun 3. PMID 23742897
- [Background] Wang P, Connor AL, Guo E, Nambao M, Chanda-Kapata P, Lambo N, Phiri C. Measuring the impact of non-monetary incentives on facility delivery in rural Zambia: a clustered randomised controlled trial. Trop Med Int Health. 2016 Apr;21(4):515-24. doi: 10.1111/tmi.12678. PMID 26848937
- [Background] WHO. Making pregnancy safer: the critical role of the skilled attendant. A joint statement by WHO, ICM, and FIGO. Geneva: Department of Reproductive Health and Research, World Health Organization. 2004.
- [Background] WHO. Making pregnancy safer the critical role of the skilled attendant: a joint statement by WHO, ICM and FIGO. Geneva: World health organization (WHO). Department of Reproductive Health and Research (RHR). 2004.
- [Derived] Mudhune S, Phiri SC, Prescott MR, McCarthy EA, Banda A, Haimbe P, Mwansa FD, Mwiche A, Silumesii A, Micheck K, Shakwelele H, Prust ML. Improving the quality of childbirth services in Zambia through introduction of the Safe Childbirth Checklist and systems-focused mentorship. PLoS One. 2020 Dec 30;15(12):e0244310. doi: 10.1371/journal.pone.0244310. eCollection 2020. PMID 33378372
- [Derived] Mudhune S, Phiri SC, Prescott MR, McCarthy EA, Banda A, Haimbe P, Mwansa FD, Mwiche A, Bwalya F, Kabamba M, Shakwelele H, Prust ML. Impact of the Safe Childbirth Checklist on health worker childbirth practices in Luapula province of Zambia: a pre-post study. BMC Public Health. 2018 Jul 18;18(1):892. doi: 10.1186/s12889-018-5813-y. PMID 30021547
- See also: Maternal mortality factsheet. Updated November 2016 — http://www.who.int/mediacentre/factsheets/fs348/en/.